CLINICAL TRIAL: NCT05395793
Title: The Role of In-person Focus Groups in the Management of Urinary Incontinence in Women From a Mixed-methods, Randomized Pilot Study
Brief Title: In-person Focus Groups in the Management of Urinary Incontinence in Women
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aqsa A. Khan, MD, Assistant Professor Department of Urology, Mayo Clinic
Other Study IDs: 18-009815
Record Dates: First submitted 2022-04-12; First posted 2022-05-27 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Self-Help Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Support Group — Support Group with moderator

SUMMARY:
The purpose of this study is to investigate how a support group with other individuals who share the condition urinary incontinence (UI) impacts patients experience with management of urinary incontinence.

DETAILED DESCRIPTION:
Focus groups in various settings have demonstrated the ability to alleviate psychological and physiological distress in focus group participants. The exploration of focus groups is warranted to measure the potential benefit for patients with urinary incontinence. Researchers aimed to assess the feasibility and acceptability of in-person focus groups as a potential intervention for female patients with urinary incontinence from a mixed methods approach. A mixed methods pilot study will be conducted to investigate whether in-person focus group demonstrate meaningful significance in quantitative outcomes measured by validated questionnaires and qualitative outcomes analyzed from focus group transcripts and post-session surveys. This study was an initial assessment to determine whether in-person focus groups for females with UI is strong enough to warrant further research and clinical implementation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* Have the ability to commute to the meeting facility without institutional assistance

Exclusion Criteria:

• Those unable to attend all three focus group sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with urinary incontinence
Study Population: Adult women with incontinence who are able to attend all three focus groups
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Change in mixed urinary incontinence symptoms | Baseline, 12 weeks
  Measured using the Medical, Epidemiological, and Social Aspects of Aging (MESA) incontinence questionnaire which consists 15 questions to measure urgency of urinary incontinence and stress urinary incontinence on a 0-3 scale (0=Never, 3=Often). Higher total scores indicating higher severity of urge and stress incontinence.
Change in urinary distress | Baseline, 12 weeks
  Measured using the Urogential Distress Inventory-6 (UDI-6) questionnaire which consists of 6 questions that rate urinary distress experience and how much it subjects are bothered by them on a 0-3 scale (0=not at all; 3=greatly).
Change in overactive bladder satisfaction with treatment | Baseline, 12 weeks
  Measured using the Overactive Bladder Satisfaction with Treatment Questionnaire (OAB-SAT-q) which consists of 11 questions rating satisfaction or dissatisfaction with treatment for overactive bladder.
Change in urinary tract condition severity | Baseline, 12 weeks
  Measured using the Patient Global Impression of Severity (PGI-S) questionnaire which consists of one question that asks subject to describe urinary tract condition currently on a scale of 1=normal, 2=mild, 3=moderate, 4=severe.
Change in urinary tract condition improvement | Baseline, 12 weeks
  Measured using the Patient Global Impression of Improvement (PGI-I) questionnaire which consists of one question that asks subject to rate urinary tract condition currently, compared with how it was before taking medication on a scale of 1-7 (1=very much better; 7=very much worse)
Change in sexual quality of life | Baseline, 12 weeks
  Measured using the Sexual Quality of Life Questionnaire- Female (SQoL-F) which consists of 18 questions to assess the relationship of sexual dysfunction and quality of life on a scale of 1-6 (1=completely agree; 6=completely disagree. Higher total scores indicate greater quality of life.
Change in Patient Health Questionnaire | Baseline, 12 weeks
  Measured using the Patient Health Questionnaire (PHQ-9) which consists of 9 questions to assess depressive symptoms using a scale of 0-3 (0=not at all; 3=nearly every day). Higher total scores indicate greater severity depression.
Change in physical activity | Baseline, 12 weeks
  Measured using the International Physical Activity Questionnaire (IPAQ) to assess physical activity as part of everyday life.

SECONDARY OUTCOMES:
Measure feasibility and acceptability of focus group | Baseline, 2 weeks, 4 weeks
  written survey was administered at the beginning of each focus group session which incorporated open-ended warm-up questions regarding urinary incontinence and concluded with the assessment of the level of focus group comfort on a scale from 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Aqsa Khan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials